CLINICAL TRIAL: NCT04281368
Title: Analysis of All Stillbirths in Stockholm County 2017, a Multidisciplinary Audit
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Wiberg-Itzel, Associate professor, Karolinska Institutet
Other Study IDs: IUFD
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Intra-Uterine Death
Keywords: IUFD
MeSH Terms: conditions — Stillbirth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analysis of IUFD — Each team member in the audit group had access to all the medical patient charts from the hospitals and also the majority of the charts from the antenatal care clinics (ANC). Each team member independently assessed each case regarding causes of death, preventable/non-preventable deaths, the level of delay if there was any and the standard of healthcare provided to the patients with stillbirth, the postmortem examination of infant and mother and if there were any recommendations given for the next pregnancy

SUMMARY:
All stillbirths in Stockholm during 2017 were analysed according to the primary outcomes which were preventable/non-preventable deaths and the level of delay. The secondary outcomes were: causes of death, standard of care pre and post stillbirth and if a summary of the possible causes of death was made as well as the planning of supervision of the next pregnancy.

DETAILED DESCRIPTION:
This is a retrospective cohort study. A multidisciplinary team consisting of three obstetricians, one midwife and one neonatologist was assembled. The team represented the largest hospitals in the region-Karolinska University Hospital and Stockholm Soderl Hospital. Each team member in the audit group had access to all the medical patient charts from the hospitals and also the majority of the charts from the antenatal care clinics (ANC). Each team member independently assessed each case regarding causes of death, preventable/non-preventable deaths, the level of delay if there was any and the standard of healthcare provided to the patients with stillbirth, the postmortem examination of infant and mother and if there were any recommendations given for the next pregnancy. Multiple meetings were organized for discussing the results of the individual assessment of each case. To enable an ethical discussion every member of the audit group signed a confidentiality form and all cases were assessed by comparison with local guidelines in praxis.

ELIGIBILITY:
Inclusion Criteria:

* All stillbirths in Stockholm 2017

Exclusion Criteria:

* Missed abortion

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: All stillbirths in Stockholm 2017
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
The rate of preventable/non-preventable deaths and the level of delay | 2017
  to analyze preventable/non-preventable deaths and the level of delay

SECONDARY OUTCOMES:
The frequency of different causes of death | 2017
  To analyze the different causes of death

CONTACTS AND LOCATIONS:
Overall Officials: Eva Wiberg-Itzel, PhD, Principal Investigator — KI
Locations (1):
- Eva Wiberg-Itzel, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sterpu I, Bolk J, Perers Oberg S, Hulthen Varli I, Wiberg Itzel E. Could a multidisciplinary regional audit identify avoidable factors and delays that contribute to stillbirths? A retrospective cohort study. BMC Pregnancy Childbirth. 2020 Nov 16;20(1):700. doi: 10.1186/s12884-020-03402-z. PMID 33198695